CLINICAL TRIAL: NCT06311526
Title: Mechanism of Action of Focal Extracorporeal Shock Waves as a Treatment of Upper Limb Stroke Spasticity: a Pilot Study
Acronym: SASHA
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 24C303
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Hemiparesis; Hemiplegia; Spasticity as Sequela of Stroke; Upper Limb Hypertonia
Keywords: Spasticity; Stroke; Extracorporeal Shockwave Therapy; Stroke upper limb impairment; Neurophysiology; Musculoskeletal ultrasound
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients suffering a spastic upper limb paresis
  Interventions: Other: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Other: Extracorporeal Shockwave Therapy — Extracorporeal Shockwave Therapy administered to the belly of spastic muscles of the upper limb.

SUMMARY:
Spasticity, common after a stroke, aggravates the patient's motor impairment causing pain and limitation in daily activities such as eating, dressing and walking.

There are different spasticity treatments, such as botulinum neurotoxin, in the first place. Among the emerging therapies is focal extracorporeal shock wave therapy, consisting of a sequence of sonic (mechanical) impulses with high peak pressure.

Systematic reviews highlighted that shock waves effectively improve lower and upper limb spasticity. Moreover, the shock waves therapeutic effect can last up to 12 weeks from the last treatment session.

When used to treat stroke spasticity, the shock waves' mechanism of action is poorly detailed.

On the one side, shock waves could change the physical properties of the muscular tissue (e.g. viscosity, rigidity).

On the other, the shock waves produce a robust mechanical stimulation that massively activates muscle and skin mechanoreceptors (e.g. muscle spindles). This activation would modulate, in turn, the spinal (and supra-spinal) circuits involved in spasticity.

To our knowledge, no study investigated the shock waves mechanism of action in stroke upper limb spasticity.

Research question: do shock waves exert their therapeutic effect on spasticity by changing the muscle's physical properties or by indirectly modulating the excitability of spinal circuits?

Specific aims: To investigate the mechanism of action of shock wave therapy as a treatment of upper limb spasticity after a stroke.

Two major hypotheses will be contrasted: shock waves reduce hypertonia 1) by changing the muscle's physical features or 2) by changing the motoneurons excitability and the excitability of the stretch reflex spinal circuits.

Shock wave therapy is expected to improve spasticity, thus improving the following clinical tests: the Modified Ashworth Scale (an ordinal score of spasticity) and the Functional Assessment for Upper Limb (FAST-UL, an ordinal score of upper limb dexterity).

This clinical improvement is expected to be associated with changes in spastic muscle echotexture assessed with ultrasounds, such as an improvement in the Heckmatt scale (an ordinal score of muscle echotexture in spasticity).

Clinical improvement is also expected to be associated with an improvement in the following neurophysiological parameters: a reduction of the H/Mmax ratio (an index of hyperexcitability of the monosynaptic stretch reflex circuit), a decrease in amplitude of the F waves (a neurophysiological signal reflecting the excitability of single/restricted motoneurones) and an increase of the homosynaptic depression (also known as post-activation depression, reflecting the excitability of the transmission between the Ia fibres and motoneurones).

Understanding the shock wave mechanism of action will lead to a better clinical application of this spasticity treatment.

If the shock waves exert their therapeutic effect by changing the muscle's physical properties, they could be more appropriate for patients with muscle fibrosis on ultrasounds.

On the contrary, if the shock waves work on spasticity by indirectly acting on the nervous system's excitability, then a neurophysiology study could be used to preliminary identify the muscle groups with the most significant neurophysiological alterations, which could be the muscles benefitting the most from this treatment.

ELIGIBILITY:
Inclusion criteria

* age > 18 years
* first hemispheric stroke at least six months ago
* spasticity of wrist and elbow flexors muscles with grade 1 to 3 of the Modified Ashworth Scal
* no botulinum toxin injection in the previous six months
* ability to give informed consent

Exclusion criteria

* anticoagulant medicine
* presence of a pacemaker, an implantable cardioverter defibrillator or other medical devices
* active cancer
* skin lesions at the site of shock wave administration
* an major neurological disease in addition to the hemiparesis (e.g. spastic hemiparesis in a patient who had Parkinson's disease before their stroke).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients with an upper limb spastic paresis.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
M wave and H reflex recruitment curve | At baseline, after 7, 14 and 21 days of intervention, at 28 and 84 days after the end of the intervention
  Recruitment curves of the Flexor Carpi Radialis muscle of both upper limbs
H reflex post-activation depression | At baseline, after 7, 14 and 21 days of intervention, at 28 and 84 days after the end of the intervention
  Post-activation depression of the Flexor Carpi Radialis H reflex of both sides
F waves | At baseline, after 7, 14 and 21 days of intervention, at 28 and 84 days after the end of the intervention
  F waves of the First Dorsal Interosseus muscles of both upper limbs
T reflex | At baseline, after 7, 14 and 21 days of intervention, at 28 and 84 days after the end of the intervention
  T reflex of the Flexor Carpi Radialis of both sides

SECONDARY OUTCOMES:
Upper limb dexterity measures | At baseline, after 7, 14 and 21 days of intervention, at 28 and 84 days after the end of the intervention
  Functional Assessment Test for Upper Limb
Ultrasound arm and forearm assessment | At baseline, after 7, 14 and 21 days of intervention, at 28 and 84 days after the end of the intervention
  Echographic assessment of the arm and forearm muscles

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The database will be made available upon request on Zenodo.

REFERENCES:
- [Background] Wissel J, Manack A, Brainin M. Toward an epidemiology of poststroke spasticity. Neurology. 2013 Jan 15;80(3 Suppl 2):S13-9. doi: 10.1212/WNL.0b013e3182762448. PMID 23319481
- [Background] Manganotti P, Amelio E. Long-term effect of shock wave therapy on upper limb hypertonia in patients affected by stroke. Stroke. 2005 Sep;36(9):1967-71. doi: 10.1161/01.STR.0000177880.06663.5c. Epub 2005 Aug 18. PMID 16109905
- [Background] Opara J, Taradaj J, Walewicz K, Rosinczuk J, Dymarek R. The Current State of Knowledge on the Clinical and Methodological Aspects of Extracorporeal Shock Waves Therapy in the Management of Post-Stroke Spasticity-Overview of 20 Years of Experiences. J Clin Med. 2021 Jan 12;10(2):261. doi: 10.3390/jcm10020261. PMID 33445623
- [Background] Pierrot-Deseilligny, E. & Burke, D. Contribution of Spinal Pathways to the Pathophysiology of Movement Disorders. The Circuitry of the Human Spinal Cord 565-579 (2012) doi:10.1017/CBO9781139026727.015.
- [Background] Kohn AF, Floeter MK, Hallett M. Presynaptic inhibition compared with homosynaptic depression as an explanation for soleus H-reflex depression in humans. Exp Brain Res. 1997 Sep;116(2):375-80. doi: 10.1007/pl00005765. PMID 9348136
- [Background] Lundbye-Jensen J, Nielsen JB. Immobilization induces changes in presynaptic control of group Ia afferents in healthy humans. J Physiol. 2008 Sep 1;586(17):4121-35. doi: 10.1113/jphysiol.2008.156547. Epub 2008 Jul 3. PMID 18599534
- [Background] Lamy JC, Wargon I, Mazevet D, Ghanim Z, Pradat-Diehl P, Katz R. Impaired efficacy of spinal presynaptic mechanisms in spastic stroke patients. Brain. 2009 Mar;132(Pt 3):734-48. doi: 10.1093/brain/awn310. Epub 2008 Nov 26. PMID 19036767